CLINICAL TRIAL: NCT00490256
Title: Evaluation of a Modified Perfusion Strategy for Neonatal Aortic Arch Reconstruction: Does Perfusing the Lower Body During Arch Repair Help?
Brief Title: Modified Perfusion for Neonatal Aortic Arch Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Brian Kogon, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002654
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Aortic Arch Hypoplasia or Atresia
Keywords: Selective Cerebral Perfusion; Renal Complications; Gastrointestinal Complications; Aortic Arch Reconstruction; Modified Perfusion; Cardiopulmonary Bypass; Pediatrics; Cardiac Defects; intestinal ischemia; necrotizing entercolitis; Near Infra-red spectroscopy; Creatinine; C-reactive protein levels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Arm 1 is the control arm. This arm will receive the standard cardiopulmonary bypass circuit.
- Experimental (Active Comparator): This arm is the modified selective perfusion arm. This arm will receive the modified cardiopulmonary circuit.
  Interventions: Procedure: Modified Selective Cerebral Perfusion

INTERVENTIONS:
Procedure: Modified Selective Cerebral Perfusion — Modified Selective perfusion is a cardiopulmonary bypass circuit that has been modified to allow blood flow to the lower body as well as the upper body while the surgery is being performed.
  Arms: Experimental

SUMMARY:
Even though the lower part of the body does receive some blood supply during Cardiopulmonary Bypass(CPB) surgery, it may not be enough. As a result of this lowered blood supply, there are complications associated with CPB and clamping of the aorta. These include complications with the stomach, intestines and kidneys.

The hypotheses of this study are that increased lower body perfusion during aortic arch reconstruction will decrease intestinal ischemia and the incidence of necrotizing enterocolitis, improve renal function in the postoperative period, and shorten both intensive care unit and hospital length of stay.

The purpose of this research study is to provide the lower part of the body and its organs with possibly more blood supply with a modified form of cardiopulmonary bypass and see if this additional blood supply helps to decrease complications of the kidney, stomach and intestines.

DETAILED DESCRIPTION:
As the aorta is repaired, the child has no circulation to the body or brain. While short periods of circulatory arrest were well tolerated, a modified technique called selective cerebral perfusion was developed to maintain blood flow to the brain during aortic repairs so as to allow for less hurried repairs with less concern over brain ischemia and injury.

Selective cerebral perfusion is designed to provide flow to the brain via the right carotid artery and collateral intracranial vessels while the aortic arch is isolated for repair. It is felt that collateral vessels also allow some perfusion of the lower body, but the adequacy of lower body perfusion during selective cerebral perfusion has not been well documented. While it is clear that some blood reaches the lower body, the incidence of renal and gastrointestinal complications following cardiac repairs involving aortic arch reconstructions remains significant.

The goal of this proposal is to evaluate a simple modification of the standard selective cerebral perfusion protocol designed to increase perfusion to the lower body during aortic arch reconstructions. Essentially all children who undergo aortic arch reconstruction at Egleston hospital have either a femoral or umbilical artery catheter in place for routine monitoring. During selective cerebral perfusion, the descending thoracic aorta is clamped, so the lower body arterial line is not a useful monitor at that point. We propose to connect a pressure line from the cardiopulmonary bypass circuit to the lower body arterial catheter, allowing for increased perfusion of the lower body through the femoral/umbilical arterial catheter during selective cerebral perfusion We will monitor simultaneous near infra-red spectroscopy of the brain, flank, and thigh to determine the adequacy of oxygen delivery to the brain, kidney, and lower body musculature during the procedure. Near infra-red spectroscopy provides a measure of the oxygenation of hemoglobin in arterial, capillary, and venous blood within the path of an infra-red sensor. Blood samples will be collected before skin incision, at the end of the procedure, and at 3, 12, and 24 hours after arrival to the intensive care unit. Intestinal fatty acid binding protein (i-FABP) and c-reactive protein (CRP) serum levels will be measured at each timepoint as markers of intestinal ischemia and generalized inflammation respectively. The incidence of documented or suspected necrotizing enterocolitis prior to hospital discharge and the time required to achieve full enteral feeds will be recorded. Renal function will be assayed by the maximal change from preoperative to postoperative serum creatinine, normalized urine output per 12 hour period following surgery, total diuretic dose per day, and daily creatinine clearance for the first 3 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis including aortic coarctation, arch hypoplasia, or interrupted aortic arch which requires cardiopulmonary bypass for repair
* age less than 1 year
* parental consent for participation

Exclusion Criteria:

* prior aortic arch operations
* emergency operation
* operating surgeon decides that selective cerebral perfusion is not indicated
* Documented renal insufficiency (creatinine > 2.0) or evidence of bowel ischemia prior to surgery

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kirshbom, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Jeffries HE, Wells WJ, Starnes VA, Wetzel RC, Moromisato DY. Gastrointestinal morbidity after Norwood palliation for hypoplastic left heart syndrome. Ann Thorac Surg. 2006 Mar;81(3):982-7. doi: 10.1016/j.athoracsur.2005.09.001. PMID 16488706
- [Background] Asou T, Kado H, Imoto Y, Shiokawa Y, Tominaga R, Kawachi Y, Yasui H. Selective cerebral perfusion technique during aortic arch repair in neonates. Ann Thorac Surg. 1996 May;61(5):1546-8. doi: 10.1016/0003-4975(96)80002-S. PMID 8633985
- [Background] Pigula FA, Siewers RD, Nemoto EM. Regional perfusion of the brain during neonatal aortic arch reconstruction. J Thorac Cardiovasc Surg. 1999 May;117(5):1023-4. doi: 10.1016/S0022-5223(99)70387-9. No abstract available. PMID 10220701
- [Background] Pigula FA, Gandhi SK, Siewers RD, Davis PJ, Webber SA, Nemoto EM. Regional low-flow perfusion provides somatic circulatory support during neonatal aortic arch surgery. Ann Thorac Surg. 2001 Aug;72(2):401-6; discussion 406-7. doi: 10.1016/s0003-4975(01)02727-8. PMID 11515874

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Experimental
Started | 7 | 7
Intraoperative Portion of the Study | 7 (Intraoperative management) | 7 (Intraoperative management)
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 7 | 14
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (8.5) | 4.7 (2.9) | 7.3 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Intestinal Fatty Acid Binding Protein and C-reactive Protein
Time Frame: Baseline and 0, 3, 12, and 24 hours after surgery
Reporting Status: Not Posted

2. Secondary Outcome: Cerebral and Lower Body Near Infra-red Spectroscopy Measures
Time Frame: 24 hours
Reporting Status: Not Posted

3. Primary Outcome: iFAB Post-op
Description: intestinal fatty acid binding protein level immediately postop
Time Frame: Immediate postop
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 7
mcg/ml | 1590 (1188) | 564 (272)

ADVERSE EVENTS:
Arm/Group | Control | Experimental
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers for analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No